CLINICAL TRIAL: NCT05664685
Title: Optimized Bismuth Quadruple Therapy vs Triple Standard Therapy for Helicobacter Pylori Eradication: Clinical Efficacy Randomized Trial
Brief Title: Optimized Bismuth Quadruple Therapy vs Triple Standard Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 220710002
Record Dates: First submitted 2022-10-08; First posted 2022-12-27 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, controlled, double-blind clinical trial with two parallel arms. The control group will receive the current Standard Triple Therapy for the eradication of H. pylori. It consists in omeprazole + amoxicillin + clarithromycin for 14 days. The intervention group will be administered Quadruple Therapy with Bismuth, that consists in esomeprazole + amoxicillin + metronidazole + bismuth subsalicylate for 14 days
Who Masked: Participant, Care Provider, Investigator
Masking Description: For the anonymization of the sequence, the research team will delegate the generation of the random sequence and the numbering of the containers to a team that has no participation or knowledge of the design of the study, the collection or analysis of data.
  The research team will deliver 204 containers with the intervention or control (102 of each) to 1 member of the UC Pharmacology and Toxicology Program. They will generate the randomization sequence, number the containers according to their result and keep the record of the randomization sequence until the data collection is finished, and the statistical analysis is done then the blind opens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will be treated with Esomeprazole 40 mg every 8 hours, Amoxicillin 1 gr every 8 hours, Metronidazole 500 mg every 8 hours, Bismuth subsalicylate 369 mg every 8 hours.
  Interventions: Drug: Optimized bismuth quadruple therapy
- Control (Active Comparator): The control group will be treated with Omeprazole 20mg every 12 hours, Amoxicillin 1 gr every 12 hours, Clarithromycin 500 mg every 12 hours, Placebo identical to Bismuth Subsalicylate, 3 times daily.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Optimized bismuth quadruple therapy — Scheme that have high dosage of amoxicillin, metronidazole and omeprazole, with bismuth. The rationale of this scheme is that in Chile, amoxicillin resistance is low, clinical metronidazole is low in the doses used and the high doses ob Proton Pump Inhibitor enhanced the antimicrobial drugs
  Other Names: Rama Intervención
  Arms: Intervention
Drug: Control — Standard eradication therapy using omeprazole, clarithromycin and amoxicillin
  Other Names: Rama Control
  Arms: Control

SUMMARY:
This study have as primary aim "To compare the H. pylori eradication rate between the quadruple bismuth therapy versus the standard triple therapy recommended by the AUGE Clinical Guidelines for Helicobacter pylori eradication treatment in peptic ulcer patients."

Briefly, this is a randomized, multicenter, controlled, double-blind clinical trial with two parallel arms. The control group will receive the current Standard Triple Therapy for the eradication of H. pylori. It consists of omeprazole + amoxicillin + clarithromycin for 14 days. The intervention group will be administered Quadruple Therapy with Bismuth, which consists in esomeprazole + amoxicillin + metronidazole + bismuth subsalicylate for 14 days

DETAILED DESCRIPTION:
Participants, all with helicobacter pylory test positive, will be recruited into the UC-CHRISTUS Health Network located in the City of Santiago de Chile for this randomized controlled clinical trial.

The intervention group will be treated with Esomeprazole 40 mg every 8 hours, Amoxicillin 1 gr every 8 hours, Metronidazole 500 mg every 8 hours, Bismuth subsalicylate 369 mg every 8 hours. The control group will be treated with Omeprazole 20mg every 12 hours, Amoxicillin 1 gr every 12 hours, Clarithromycin 500 mg every 12 hours, Placebo identical to Bismuth Subsalicylate, 3 times daily.

The primary outcome is H. pylori Eradication. To determine eradication, participants of these study will be invited 8 to 12 weeks after the end of the administered therapy.

As secondary outcomes, will be recorded the Incidence of Adverse Drug Reactions (ADRs) through a questionnaire that will be performed to determine the occurrence of any adverse effect attributable to the therapy. The incidence of bloating, abdominal pain, bitter taste, constipation, diarrhea, dizziness, dyspepsia, epigastric pain, halitosis, headache, loss of appetite, nausea, vomiting, oral ulcers, skin rashes, and drowsiness will be directly recorded. Symptoms reported by participants spontaneously in follow-up phone calls will also be recorded. The time of commencement and duration of the therapy will be recorded. Also will be measured the H. pylori Antibiotic Resistance and Host CYP2C19 polymorphisms determination.

Covariates will be recorded at recruitment. For ADRs and therapeutic adherence telephone follow-up will be performed on days 7 and 14 and 21 after initiation of the therapy. The last follow-up will be performed in person at the time of the UBT.

Sample size calculation

For sample size calculations the following are considered: the expected Eradication rate with the control therapy scheme 82%, the expected eradication rate with the intervention therapy scheme: 97%, the expected absolute difference between therapies 15%, Power 80%, and confidence 95%

This calculation results that 65 participants per branch are needed. Calculations were performed with the statistical program Stata 15. Considering a loss of 10.0%, 72 patients per branch are considered. In addition, the investigators considered 30 additional patients in case the groups resulting from randomization are not balanced, and it is necessary to adjust the effectiveness of the treatments, by 3 variables to be able to make a regression analysis. With this, a total of 102 patients per branch will be included in this study.

Methods used to generate the sequence for patient random assignment to branches For the assignment of participants in the intervention or control branches, a list of random numbers will be used to sequence containers containing the control or intervention treatments. The containers will be delivered to the study participants according to the order in which participants are recruited.

The mechanism used to implement branch random assignment

For the anonymization of the sequence, the research team will delegate the generation of the random sequence and the numbering of the containers to a team that has no participation or knowledge of the design of the study, the collection, or the analysis of data.

Generation of the assignment sequence, recruitment of participants, and assignment of participants to the intervention's responsibilities.

The research team will deliver 204 containers with the intervention or control (102 of each) to 1 member of the UC Pharmacology and Toxicology Program. The member will generate the randomization sequence, number the containers according to their result, and keep the record of the randomization sequence until the data collection is finished, and the statistical analysis is done then the blind opens. In this way responsibilities are assigned to:

A. Generation of the branch assignment sequence: UC Pharmacology and Toxicology Program B. Participant Recruitment: Principal Investigator C. Assignment of participants to the interventions: Principal investigator delivers the containers to the participants, keeping them blind by the randomization and previous numbering of the containers.

Blind status maintenance for participants and research team

To maintain a blind status to branch assignment:

A. Part of the research team that performs patients recruitment B. Part of the research team that performs follows up on participants C. Part of the research team that performs tests for confirmation of eradication of H. pylori D. Part of the research team that performs statistical analysis

Statistical methods used for group comparison of primary and secondary outcomes

The statistical analysis will be performed without knowledge of the therapy scheme assignment, or the clinical evaluation of participants included in the study. P values <0,05 will be considered statistically significant. The analyses will be carried out under the intention-to-treat (ITT) modality.

Registration and safeguarding of the data collected

Data logging has 3 stages:

1. Recruitment
2. Telephone follow-ups on days 7, 14, and 21 after starting treatment.
3. UBT exam between 8 and 12 weeks after treatment ends.

Each stage will have a physical record on paper, which will be transcribed into the REDCap electronic registry. The paper records will be maintained under lock and key at the Toxicological and Drug Information Center (CITUC), located at Lira 63, second floor.

Regarding the quality of the data recorded

At the time of analysis, a random sample of 10% of the participants will be selected to evaluate the consistency between the physical and electronic records. If there are doubts about the quality of the information, all records will be checked. Anomalous values will also be checked in the physical register.

Data Analysis Plan

Descriptive Statistics

Descriptive statistics will be performed to determine the characteristics of the complete cohort and stratified by experimental branch. The balance of the intervention and control groups will be evaluated. If the balance is not reached, the effect will be directly adjusted with multivariate models.

Primary analysis: Comparison of treatment efficacy

The analysis will perform a comparison of eradication percentages between groups by inferential statistical tests, to determine whether the difference between the groups reaches statistical significance, and also calculate relative risk measures. There will be analyzed variables associated with positive eradication and multivariate analysis of factors associated with eradication using binomial regression.

Secondary analysis: Adverse drug reactions

Adverse reactions

Will be performed descriptive statistics, by type, particular symptom, and temporal evolution. Comparison between control and intervention branches will be analyzed by the magnitude of ADR observed. Evaluation of the association between ADR s with treatment scheme and covariates, by regression, will be performed.

Sensitivity analysis

To evaluate the robustness of the results, the analysis will be repeated in the modality by protocol to compare them with those obtained under the intention-to-treat modality. Secondly, the effect of therapeutic adherence will be evaluated. The analysis will also be stratified by the measured covariates, to evaluate sources of uncertainty, confusion, or possible interactions.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with H. pylori infection by positive Urease test.

Exclusion Criteria:

* Pregnant or lactating women.
* Allergy or history of adverse reaction to the following medications:
* Penicillin
* Salicylate allergy
* Omeprazole
* Has received H. pylori eradication therapy prior to the study.
* Has used PPIs 14 day prior to diagnostic testing
* Use of antibiotics within 4 weeks beforehand.
* History of gastrointestinal bleeding for the last 12 weeks.
* History of partial gastrectomy due to Gastric Cancer
* History of incipient Gastric Cancer resolved by endoscopic resection.
* History of bariatric surgery.
* Serious or malignant diseases with less than 1 year life expectancy.
* History of Clostridium difficile infection.
* History of inflammatory bowel disease.
* Chronic kidney disease, stage 3 or higher.
* Do not sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori erradication | 8-12 weeks after treatment is ended
  Determined by Urea breath test for Helicobacter pylori

SECONDARY OUTCOMES:
Incidence of Adverse Drug Reactions | Day 7, 14 and 21 after treatment begins
  A questionnaire will be performed to determine the occurrence of any adverse effect attributable to the therapy
Prevalence of Helicobacter pylori antibiotic resistance to Clarithromycin | Samples taken at the recruitment
  To determine the susceptibility to Clarithromycin, PCRs will be performed with specific allele primers (ASP-PCR) for point mutations A2142G and A2143G of the H. pylori 23s rRNA gene
Prevalence of Host CYP2C19 polymorphisms determination | Samples taken at the recruitment
  To perform host CYP2C19 polymorphisms genotyping real time PCR using TaqMan probes for the Drug Metabolism Genotyping Assay of the to detect variants *2 (c.681G >A; rs 4244285), *3 (c. 636G >A; RS 4986893) and *17 (-806C >T; RS 12248560).

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Medel, MPH, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (2):
- Chile (2):
  - Centro de especialidades médicas Marcoleta UC CHRISTUS, Santiago, Santiago Metropolitan
  - Centro Médico UC-CHRISTUS San Joaquín, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FitzGerald R, Smith SM. An Overview of Helicobacter pylori Infection. Methods Mol Biol. 2021;2283:1-14. doi: 10.1007/978-1-0716-1302-3_1. PMID 33765303
- [Background] McColl KE. Clinical practice. Helicobacter pylori infection. N Engl J Med. 2010 Apr 29;362(17):1597-604. doi: 10.1056/NEJMcp1001110. No abstract available. PMID 20427808
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Rollan A, Arab JP, Camargo MC, Candia R, Harris P, Ferreccio C, Rabkin CS, Gana JC, Cortes P, Herrero R, Duran L, Garcia A, Toledo C, Espino A, Lustig N, Sarfatis A, Figueroa C, Torres J, Riquelme A. Management of Helicobacter pylori infection in Latin America: a Delphi technique-based consensus. World J Gastroenterol. 2014 Aug 21;20(31):10969-83. doi: 10.3748/wjg.v20.i31.10969. PMID 25152601
- [Background] Ferreccio C, Rollan A, Harris PR, Serrano C, Gederlini A, Margozzini P, Gonzalez C, Aguilera X, Venegas A, Jara A. Gastric cancer is related to early Helicobacter pylori infection in a high-prevalence country. Cancer Epidemiol Biomarkers Prev. 2007 Apr;16(4):662-7. doi: 10.1158/1055-9965.EPI-06-0514. PMID 17416755
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Background] Chiang TH, Chang WJ, Chen SL, Yen AM, Fann JC, Chiu SY, Chen YR, Chuang SL, Shieh CF, Liu CY, Chiu HM, Chiang H, Shun CT, Lin MW, Wu MS, Lin JT, Chan CC, Graham DY, Chen HH, Lee YC. Mass eradication of Helicobacter pylori to reduce gastric cancer incidence and mortality: a long-term cohort study on Matsu Islands. Gut. 2021 Feb;70(2):243-250. doi: 10.1136/gutjnl-2020-322200. Epub 2020 Aug 13. PMID 32792335
- [Background] Greenberg ER, Anderson GL, Morgan DR, Torres J, Chey WD, Bravo LE, Dominguez RL, Ferreccio C, Herrero R, Lazcano-Ponce EC, Meza-Montenegro MM, Pena R, Pena EM, Salazar-Martinez E, Correa P, Martinez ME, Valdivieso M, Goodman GE, Crowley JJ, Baker LH. 14-day triple, 5-day concomitant, and 10-day sequential therapies for Helicobacter pylori infection in seven Latin American sites: a randomised trial. Lancet. 2011 Aug 6;378(9790):507-14. doi: 10.1016/S0140-6736(11)60825-8. Epub 2011 Jul 21. PMID 21777974
- [Background] Tshibangu-Kabamba E, Yamaoka Y. Helicobacter pylori infection and antibiotic resistance - from biology to clinical implications. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):613-629. doi: 10.1038/s41575-021-00449-x. Epub 2021 May 17. PMID 34002081
- [Background] Ierardi E, Losurdo G, Fortezza RF, Principi M, Barone M, Leo AD. Optimizing proton pump inhibitors in Helicobacter pylori treatment: Old and new tricks to improve effectiveness. World J Gastroenterol. 2019 Sep 14;25(34):5097-5104. doi: 10.3748/wjg.v25.i34.5097. PMID 31558859
- [Background] Kuo CH, Lu CY, Shih HY, Liu CJ, Wu MC, Hu HM, Hsu WH, Yu FJ, Wu DC, Kuo FC. CYP2C19 polymorphism influences Helicobacter pylori eradication. World J Gastroenterol. 2014 Nov 21;20(43):16029-36. doi: 10.3748/wjg.v20.i43.16029. PMID 25473155
- [Background] Fallone CA, Chiba N, van Zanten SV, Fischbach L, Gisbert JP, Hunt RH, Jones NL, Render C, Leontiadis GI, Moayyedi P, Marshall JK. The Toronto Consensus for the Treatment of Helicobacter pylori Infection in Adults. Gastroenterology. 2016 Jul;151(1):51-69.e14. doi: 10.1053/j.gastro.2016.04.006. Epub 2016 Apr 19. PMID 27102658
- [Background] Arenas A, Serrano C, Quinones L, Harris P, Sandoval M, Lavanderos M, Sepulveda R, Maquilon S, Echeverria A, Rios C, Fuentes-Lopez E, Rojas L, Jorquera A, Pizarro M, Camargo MC, Riquelme A. High prevalence of clarithromycin resistance and effect on Helicobacter pylori eradication in a population from Santiago, Chile: cohort study and meta-analysis. Sci Rep. 2019 Dec 27;9(1):20070. doi: 10.1038/s41598-019-56399-7. PMID 31882676
- [Background] Gonzalez-Hormazabal P, Arenas A, Serrano C, Pizarro M, Fuentes-Lopez E, Arnold J, Berger Z, Musleh M, Valladares H, Lanzarini E, Jara L, Castro VG, Camargo MC, Riquelme A. Prevalence of Helicobacter pylori Antimicrobial Resistance Among Chilean Patients. Arch Med Res. 2021 Jul;52(5):529-534. doi: 10.1016/j.arcmed.2021.01.011. Epub 2021 Feb 12. PMID 33583603
- [Background] Camargo MC, Garcia A, Riquelme A, Otero W, Camargo CA, Hernandez-Garcia T, Candia R, Bruce MG, Rabkin CS. The problem of Helicobacter pylori resistance to antibiotics: a systematic review in Latin America. Am J Gastroenterol. 2014 Apr;109(4):485-95. doi: 10.1038/ajg.2014.24. Epub 2014 Mar 4. PMID 24589670
- [Background] Reyes D, Ortiz J, Fuentes-Lopez E, Budnik S, Gandara V, Gallardo A, Seydewitz MF, Candia R, Vargas JI, Rollan MP, Godoy J, Rollan A, Mansilla R, Arenas A, Chahuan J, Espino A, Pizarro M, Riquelme A. Quadruple therapies are superior to standard triple therapy for Helicobacter pylori first-line eradication in Chile. Gastroenterol Hepatol. 2022 Aug-Sep;45(7):515-523. doi: 10.1016/j.gastrohep.2021.11.010. Epub 2021 Dec 7. English, Spanish. PMID 34890721
- [Background] Kita T, Tanigawara Y, Aoyama N, Hohda T, Saijoh Y, Komada F, Sakaeda T, Okumura K, Sakai T, Kasuga M. CYP2C19 genotype related effect of omeprazole on intragastric pH and antimicrobial stability. Pharm Res. 2001 May;18(5):615-21. doi: 10.1023/a:1011025125163. PMID 11465416
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Valencia-Monsalvez F, Mendoza-Parra S, Luengo-Machuca L. [Evaluation of Morisky medication adherence scale (mmas-8) in older adults of a primary health care center in Chile]. Rev Peru Med Exp Salud Publica. 2017 Apr-Jun;34(2):245-249. doi: 10.17843/rpmesp.2017.342.2206. Spanish. PMID 29177383
- [Derived] Medel-Jara PA, Latorre G, Fuentes-Lopez E, Pizarro M, Viviani P, Chahuan J, Maquilon S, Corsi O, Reyes D, Espino A, Vargas JI, Wichmann IA, Harris P, Serrano C, Buruato I, Sandoval C, Varela NM, Cerpa L, Quinones L, Megraud F, Huang RJ, Shah SC, Perez AR. Comparison between optimized bismuth quadruple therapy and standard clarithromycin-based triple therapy for first-line Helicobacter pylori eradication: a double-blind randomized controlled trial. Lancet Reg Health Am. 2025 Nov 22;53:101312. doi: 10.1016/j.lana.2025.101312. eCollection 2026 Jan. PMID 41362749

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT05664685/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT05664685/ICF_001.pdf